CLINICAL TRIAL: NCT04222686
Title: Rationale and Design of a Simple Randomized Trial Evaluating Losartan and Perindopril in Blacks Type 2 Diabetics Patients: the Cardiac and Renal Protection With Losartan or Perindopril (CARE-PLP) Trial
Brief Title: Evaluation of Losartan and Perindopril in Blacks Type 2 Diabetics Patients
Acronym: CARE-PLP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CARE-PLP
Record Dates: First submitted 2019-04-08; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Angiotensin Converting Enzymes Inhibitor; Angiotensin II Receptor Blockers; Type 2 Diabetes; Exercise induced urinary albumin excretion; Blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Viacoram; Perindopril; Losartan

STUDY DESIGN:
Intervention Model Description: CARE-PLP trial is a double blind, randomized, controlled parallel clinical trial conducted in the National Obesity Center, Yaounde, Cameroon
Who Masked: Participant, Investigator
Masking Description: The double-blind model is applied to the study. Only the adjudicator, responsible for the distribution of medication knew the different regimes. Perindopril and Losartan were packaged in boxes of identical appearance and labeled for each participant by name and number of the randomization program. The randomization and packaging of the drugs was done by an investigator who had no clinical involvement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perindopril Arm (Active Comparator): 10 mg Perindopril tablet per day at 8am (+/- 1 hour) was add to the usual treatment for each patient. Patients are followed-up for a period of 08 weeks.
  Interventions: Drug: Perindopril Arginine
- Losartan Arm (Active Comparator): 100 mg Losartan tablet per day at 8am (+/- 1 hour) was add to the usual treatment for each patient. Patients are followed-up for a period of 08 weeks.
  Interventions: Drug: Losartan Potassium

INTERVENTIONS:
Drug: Perindopril Arginine — 10 mg Perindopril tablet / day will be added to the usual treatment for each patient for a period of 8 weeks.
  Other Names: Perindopril
  Arms: Perindopril Arm
Drug: Losartan Potassium — 100 mg Losartan tablet will be added to the usual treatment for each patient for a period of 08 weeks.
  Other Names: Losartan
  Arms: Losartan Arm

SUMMARY:
The aim of this study is to compare the short-term effects of ACEi and angiotensin II receptor blockers on cardiac and renal protection in black type 2 diabetics patients CARE-PLP is a double-arm, double-blind, randomized and parallel clinical trial conducted at the National Obesity Center in the Yaoundé Central Hospital. A population of Type 2 diabetes patients, with hypertension and / or microalbuminuria and who are not taking ACEi or angiotensin receptors blockers, is randomize into two groups. Depending on the group, 10 mg Perindopril or 100 mg Losartan is add to the usual treatment for each patient. The patients are followed-up for a period of 08 weeks. The primary outcome is the variation of exercise induced urinary albumin excretion after 08 weeks of intervention.

DETAILED DESCRIPTION:
Given the particularity of the renin-angiotensin system in black subjects, the CARE-PLP study fulfills this objective with the comparison of Losartan and Perindopril after 08 weeks of administration in a subsaharan African population.

Aim: The aim of this study is to compare the short-term effects of ACEi and angiotensin II receptor blockers on cardiac and renal protection in black type 2 diabetics patients

Methods: CARE-PLP is a double-arm, double-blind, randomized and parallel clinical trial conducted at the National Obesity Center in the Yaoundé Central Hospital. A population of Type 2 diabetes patients, with hypertension and / or microalbuminuria and who are not taking ACEi or angiotensin receptors blockers, is randomize into two groups. Depending on the group, 10 mg Perindopril or 100 mg Losartan is add to the usual treatment for each patient. The patients are followed-up for a period of 08 weeks. The primary outcome is the variation of exercise induced urinary albumin excretion after 08 weeks of intervention.

Progress: Recruitment for CARE-PLP was completed in february 2018 with 29 patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetics subjects
* Urinary albumin excretion >30 g/day or Blood pressure > 140/90
* On a stable antidiabetic and antihypertensive therapies (determined by the investigator) for at least 3 months with no classes changes. The pharmacological treatment should not include an angiotensin-converting enzyme inhibitor or angiotensin II receptor blocker
* Subject must not present any contraindication to exercise
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Side effects affecting life quality of patients (determined by the Data Safety Monitoring Board).
* Signs of exercise intolerance
* Out of sight.
* Withdrawal of consent

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Variation of exercise-induced urinary albumin excretion | 8 weeks
  Variation of exercise-induced urinary albumin excretion (mg/j) between week 0 and week 8. By nephelometry method.

SECONDARY OUTCOMES:
Change in rest urinary albumin excretion | 8 weeks
  Change in rest urinary albumin excretion (mg/l) from baseline to week 08. By nephelometry method.
Change in mitral E/Ea ratio | 8 weeks
  Change in mitral E/Ea ratio from baseline to week 08. By tissue doppler on echocardiography.
Change in nycthemeral blood pressure profile (mmHg) | 8 weeks
  Change in nycthemeral blood pressure profile from baseline to week 08. By using Arterial Blood Pressure Monitoring.
Change in concentration of antioxidants markers (micromol) | 8 weeks
  Change in concentration of antioxidants markers from baseline to week 08. By spectrophotometer
Change in lipid profile (triglycerides, Total cholesterol, HDL-cholesterol, LDL-cholesterol) on g/l | 8 weeks
  Change in lipid profile from baseline to week 08. By spectrophotometer
Change in uricemia concentration | 8 weeks
  Change in uricemia concentration (mg/l) from baseline to week 08. By spectrophotometer

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nadege NGANOU-GNINDJIO, MD, MAS, Principal Investigator — Yaounde Central Hospital
Locations (1):
- Yaounde Central Hospital, NAtional Obesity Center, Yaoundé, Cameroon